CLINICAL TRIAL: NCT03663374
Title: International Multicentre Randomized Double-blind Placebo Controlled Phase III Clinical Study to Assess Efficacy and Safety of Odelepran, 125 mg, for the Use in Patient With Alcohol Dependence
Brief Title: Efficacy and Safety Evaluating Study of Odelepran for the Use in Patient With Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Synergy Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN07006005
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; abstinence; alcohol abuse; LY2196044; ondelopran
MeSH Terms: conditions — Alcoholism | interventions — LY2196044

STUDY DESIGN:
Intervention Model Description: All eligible patients were randomized into two groups to receive investigational drug or placebo at ratio 1:1
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Odelepan (Experimental): One tablet once daily
  Interventions: Drug: Odelepan
- Placebo (Placebo Comparator): One tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Odelepan — Tablets, 125 mg
  Other Names: Ondelopran; LY2196044
  Arms: Odelepan
Drug: Placebo — Contains the same excipients as Odelepran but it does not contain the active agent. Placebo is identical to Odelepran in terms of drug form and external characteristics (colour, smell, etc). Doses and route of administration are identical to those for Odelepran.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess efficacy and safety of the study drug Odelepran, 125 mg as compared to placebo in the treatment of alcohol dependence in adult outpatients.

DETAILED DESCRIPTION:
Patients for this study were recruited in specialized psychiatric and addictology clinical sites in Russia and Kazakhstan. Eligible patients were randomly allocated in one of the following treatment groups in 1:1 ratio:

* The main group was taking the study drug Odelepran, one 125 mg tablet per day;
* The comparison group was taking the comparison drug (Placebo) orally, one tablet per day.

Duration of the study treatment period was 24 weeks (starting from the Day 1). Patients were keeping a diary to register their drug taking and amount and kind of alcohol beverages consumed.

Patients were not allowed to participate in psychotherapy or take any psychotropic drugs except for short-acting benzodiazepines for insomnia. However benzodiazepines were not allowed for taking less than 24 before any study visit.

Patients visited clinical sites regularly as per the Schedule for visits and procedures. During the visits to the site the patient's mental state examination with the use of psychometric scales was conducted and the study drug was provided.

Starting at randomization and subsequently at all scheduled visits investigators conducted a brief (15 minutes or less) psychotherapeutic intervention (individual counseling) during which patients were asked to provide information on aspects of alcohol consumption and emotional states experienced while abstaining from alcohol. Such individual counseling was aimed to reinforce lifestyle changes, motivate sobriety and enhance protocol adherence. All clinical sites performed such counseling in standardized manner in accordance with protocol-specific Guideline developed at St. Petersburg Psychoneurological Research Institute named after V.M. Bekhterev for the purposes of this study.28 days after the last dose of study drug patients were asked to come for a follow up visit to assess adverse events.

Patients were not paid for participation in the study.

Assessments of efficacy and safety were performed monthly. Assessments of drinking behavior were based on the Time Line Follow-Back (TLFB) method used to provide information of daily number of standard drinks. At every visit patients reported about dynamics of drinking (frequency and amount of consumed alcohol) since the previous visit.

For all assessed variables, the baseline was defined as an assessment at the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Outpatients (not hospitalized by the moment of randomization).
* Average alcohol consumption during 30 days prior to screening higher than a medium drinking risk level (men: > 4 drinks/day or 14 drinks/week; women > 3 drinks/day or 7 drinks/week) according to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria.
* Patients diagnosed with alcohol dependence according to the International Classification of Diseases (ICD)-10, assessed with the Mini-International Neuropsychiatric Interview (MINI).
* Abstaining from alcohol during 3 days prior to screening and 3 days before randomization confirmed by the test for alcohol in exhaled air (less than 0,02 %).
* For women retaining childbearing potential - negative pregnancy test and consent to use reliable contraception methods (as well as for men) throughout the study period, including the study follow up period.
* Patients able to comply with study protocol as per investigator's opinion.
* Availability of a patient's trustee who reside with the patient. A trustee is defined here as a person who spends with the patient at least 4 hours a day. The trustee must give his/her consent for participation in the study as the patient's representative.
* Study drug monotherapy must be acceptable for the patient as per investigator's opinion.

Exclusion Criteria:

* Hypersensitivity to Odelepran or to any excipient of the study drug (including lactose intolerance).
* Binge drinking (more than 5 day consecutive days of heavy drinking) during 30 days prior to screening. Heavy drinking is considered as 5 or more drinks per day for men and 4 or more drinks per day for women.
* Ever diagnosed schizophrenia, schizoaffective disorder, bipolar mood disorder or any other psychiatric disorder, except for alcohol dependence. History of alcohol induced psychosis.
* Anxiety or depressive disorder present at enrollment into the study. Montgomery-Asberg Depression Rating Scale (MADRS) score higher than 15.
* High suicidal risk confirmed by MINI.
* Previous use of opioid antagonists implants less than 3 months prior to screening; use of long-acting naltrexone injections (e,g, Vivitrol) less than 4 weeks after the first injection and 3 months after the second and the following injections; use of cyanamide (Kolme) less than 2 weeks prior to screening, use of oral opioid antagonists or disulfiram during 2 weeks prior to screening.
* Psychotherapeutic "coding" (a method when the patient is induced a misbelief that alcohol consumption would lead to death, expected to result from undisclosed pharmacological manipulation) that took place during less than 3 months prior to screening.
* Use of psychotropic medication less than 3 weeks before the screening (for long-acting and 'depot' formulations) or 1 week before the screening (for other formulations) except for those used to treat alcohol withdrawal syndrome.
* Severe alcohol withdrawal syndrome (severity of alcohol withdrawal more than 10 on Clinical Institute Withdrawal Assessment of Alcohol (CIWA-Ar) scale).
* History of seizures (excepting febrile seizers). Severe brain injury, history of intracranial neoplasms and/or intracranial haemorrhages or any conditions that impose the risk of seizures. History of anticonvulsive therapy.
* Any clinical condition affecting cognitive or other psychoneurological functioning (verified for head injury with the loss of consciousness that lasted more than 1 hour, or resulted in cognitive or behavioral impairment, stroke, encephalopathy, dementia, neurodegenerative disorder, etc). Except for mild cognitive impairment.
* Mental retardation of syndromes of severe organic brain injury.
* Use of drugs of abuse (opioids, cannabinoids, amphetamines, etc.) or diagnoses of substance addiction/dependence at the moment of screening or positive urine drug screen test.
* Significant liver function impairment (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) higher than 3 upper limits of normal range or diagnosis of hepatic failure, class B or C by Child Pugh).
* Severe renal failure (creatinine clearance calculated at the screening less than 30 ml/min or renal replacement therapy).
* Severe cardiovascular system disorders: unstable angina, poorly controlled arrhythmia, cardiac failure of III or IV class by New-York Heart Association (NYHA), acute myocardial infarction within the past 6 months.
* HIV-infection, hepatitis B or C.
* Decompensated diabetes mellitus (determined glycated hemoglobin HbAc1 level more than 7,5%)
* Other concomitant disorders and conditions that, as per investigator's opinion, put the patient's safety under risk or that could affect the analysis of safety data.
* Any diagnosed or suspected malignancy.
* Pregnancy, breast feeding.
* Participation in any other clinical study during 30 days or 6 periods of half life (depending on what is longer) prior to screening.
* Patients that need treatment with drugs prohibited by the study protocol (opioid antagonists, psychotropic medications, opioid analgesics, anticonvulsants, central muscle relaxants, antineoplastic drugs, glucocorticoids).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2016-04-16 (Actual); Study Completion 2016-05-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean daily alcohol consumption | Baseline and Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 of treatment
  Calculated as total number of drinks in month divided by number of days in month.

SECONDARY OUTCOMES:
Change in the number of days of abstinence per month as compared to the baseline | Baseline and Week 24 of treatment
Change in the percentage of days of heavy drinking per month as compared to the baseline | Baseline and Week 24 of treatment
  Heavy drinking to be considered as 5 or more drinks per day for men and 4 or more drinks per day for women.
Time to the first day of drinking | From baseline till the first day of alcohol consumption
  Full abstinence period duration.
Time to the first day of heavy drinking | From baseline till the first day of heavy drinking
  Heavy drinking to be considered as 5 or more drinks per day for men and 4 or more drinks per day for women.
Change from baseline in alcohol consumption per drinking day | Baseline and Week Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20 and 24 of treatment
  Calculated as total number of drinks in month divided by number of drinking days in month.
Change in alcohol craving from the baseline (based on Obsessive-Compulsive Drinking Scale (OCDS) score) | Baseline and Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 of treatment
  The OCDS is a validated scale consisted of 14 items for patient self-assessment of alcohol craving. Scoring by simple addition. Higher scores indicate greater level of craving (Anton R.F., Moak D.H., Latham P.K., 1996).
Change in alcohol craving (based on completed VIsual Analogue Scale) | Baseline and Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 of treatment
  VIsual Analogue Scale (VAS) ranged from 0 to 100, where 0 corresponds to "no craving at all" and 100 corresponds to "maximal craving"
Change in patient's self-assessed quality of life (by the SF-36 Questionnaire) as compared to the baseline | Baseline and Week 8, 24 of treatment
  The Short Form Health Survey (SF-36) is a validated 36 item self-report Quality of Life Questionnaire that measures eight multi-item dimensions of health: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain, and general health perception. Version 2 was used. (Ware J.E., 2000)
Proportion of patient with clinical improvement as assessed by Clinical Global Impression-improvement (CGI-I) scale | Week 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 of treatment
  CGI-I scale is a 7 point scale that requires the investigator to assess how much the patient's illness has improved or worsened relative to a baseline. Rated as: 1 - very much improved, 2 - much improved, 3 - minimally improved, 4 - no change, 5 - minimally worse, 6 - much worse, 7 - very much worse. (Guy W, 1970; 1976)
Efficacy index of CGI | Week 12 and 24 of treatment
  Efficacy index is a 4×4 rating scale that assesses the therapeutic effect of treatment with psychiatric medication (with possible considerations: 1 - unchanged or worse; 2 - minimal - slight improvement which doesn't alter status of care of patient; 3 - moderate marked - decided improvement, partial remission of symptoms; 4 - marked - vast improvement, complete or nearly complete remission of all symptoms) and associated side effects (with possible considerations: 1 - none; 2 - do not significantly interfere with patient's functioning; 3 - significantly interfere with patient's functioning; 4 - outweigh therapeutic effect). Derived by dividing therapeutic effect score by side effects score. The lower efficacy index corresponds to the better result (Guy W, 1970; 1976)
Change from baseline in the Drinker Inventory of Consequences questionnaire (DrInC-2R) total score | 3 previous months, baseline and Week 4, 8, 12, 16, 20 and 24 of treatment
  DrInC-2R is a validated self-report questionnaire consisted of 50 questions to measure adverse consequences of alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal as well as frequency of these consequences (answers given on frequency scale grade from 0-3: 0 - never, 1 - once or a few times, 2 - once or twice a week 3 - daily or almost daily). Higher scores indicate greater levels of alcohol-related problems. (Miller W.R., 1995)
Change in impulsivity (Barratt impulsivity scale by the subscales and by the total score) from the baseline | Baseline and Week 8, 16 and 24 of treatment
  Barratt impulsivity scale (BIS-11) is a validated self-report questionnaire composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Items are scored on a 4-point scale: Rarely/Never = 1, Occasionally = 2, Often = 3, Almost Always/Always = 4. Total score is assessed. The higher total score corresponds to the more impulsive behavior (Patton et al., 1995)
Proportion of patients completed the trial | Week 24 of treatment
Time to untimely withdrawal from the study | From baseline to Week 24 of treatment
Number of the early dropouts from the study | Week 24 of treatment
  Per reasons

OTHER OUTCOMES:
Number of hospitalizations due to alcohol intoxication | 6 month prior to the baseline and week 28 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (22):
- Republican Research center of psychiatry, psychotherapy and addictology, Almaty, Kazakhstan
- Russia (21):
  - Republican clinical mental hospital n.a. V.M. Bekhterev, Kazan'
  - First Moscow State Medical University named after I.M.Sechenov, Moscow
  - Institute of mental health and addictology, LCC, Moscow
  - Murmansk regional narcological dispensary, Murmansk
  - Clinical mental hospital #1, Dispensery department, Nizhny Novgorod
  - Clinical mental hospital #1,Medico-rehabilitational department, Nizhny Novgorod
  - Research center Feniks, LLC, Rostov-on-Don
  - Baltic Medicine LLC, Saint Petersburg
  - City addiction clinic, 2nd department, Saint Petersburg
  - City addiction clinic, Petrogradsky region, Saint Petersburg
  - City addiction clinic, Vasileostrovsky region, Saint Petersburg
  - Doctor SAN, LLC, Saint Petersburg
  - Eco-Safety Research Center, Saint Petersburg
  - Pavlov First Saint Petersburg State, Saint Petersburg
  - Saint Petersburg regional narcological dispensary, Saint Petersburg
  - St.Petersburg V.M. Bekhterev Psychoneurological Research Institute, addictive pathology department, Saint Petersburg
  - St.Petersburg V.M. Bekhterev Psychoneurological Research Institute, alcohol dependance department, Saint Petersburg
  - Clinical city hospital #2 n.a. V.I. Razumovsky, Saratov
  - Mental Health Research Institute, Tomsk
  - Lion-Med, LLC, Voronezh
  - Yaroslavl Region Clinical Mental Hospital, Yaroslavl

REFERENCES:
- [Background] Sobell L.C., Sobell M.B. (1992) Timeline Follow-Back. In: Litten R.Z., Allen J.P. (eds) Measuring Alcohol Consumption. Humana Press, Totowa, NJ